CLINICAL TRIAL: NCT01346553
Title: Safety and Primary Efficacy of the External Synchronized Vein Valve (ESVV) in Treatment of Chronic Venous Insufficiency (CVI) Sequel - A Pilot Study
Brief Title: Safety and Efficacy of the External Synchronized Vein Valve (ESVV) in Treatment of Chronic Venous Insufficiency (CVI)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: GB-Veintech (Industry)
Responsible Party: Dr. Hanna levy, GB-Veintech
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESVV - PS-01
Record Dates: First submitted 2011-04-30; First posted 2011-05-03 (Estimated); Last update posted 2011-05-03 (Estimated); Status verified 2011-04

CONDITIONS: Venous Insufficiency
Keywords: Chronic Venous Insufficiency (CVI)
MeSH Terms: conditions — Venous Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ESVV treatment (Experimental): using ESVV device
  Interventions: Device: ESVV device

INTERVENTIONS:
Device: ESVV device — wearing the ESVV device for 6 hours
  Other Names: Chronic Venous Insufficiency (CVI)treatment

SUMMARY:
The External Synchronized Vein Valve (ESVV), is intended for the treatment of Chronic Venous Insufficiency (CVI), incorporates an external apparatus that is aimed to replace the one-way venous valve and a sensor that identifies the movement of the calf muscles pump. The external device is located above the failed deep vein and exerts synchronized intermittent regulated pressure on it. Alteration in the vein structure is occurred and the blood flows in the cephalad direction, preventing the return toward the feet. The device is synchronized with the calf muscles pump to function as a one-way venous valve. This study was design in order to assess safety and efficacy of using the ESVV for treatment of consequences of deep chronic venous insufficiency.

ELIGIBILITY:
Inclusion Criteria:

* Males and females age 18 and up.
* Patient is diagnosed to have deep chronic venous insufficiency (CVI) proved by recent duplex examination.
* Patient able to comprehend and give informed consent for participation in this study.
* Patient must commit to both screening and treatment visits.
* Patient must sign the Informed Consent Form.

Exclusion Criteria:

* Acute deep vein thrombosis.
* Chronic deep vein obstruction.
* Peripheral arterial occlusive disease.
* Ankle edema that is not caused by chronic venous insufficiency
* Partial or complete immobility.
* Pregnancy.
* Known cognitive disorder.
* Drug abuse.
* Patient objects to the study protocol.
* Concurrent participation in any other clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2011-06; Primary Completion 2011-12 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
The safety of using the ESVV for CVI treatment | 6 hours
  Adverse events will be documented

SECONDARY OUTCOMES:
Assessing the efficacy of using the ESVV for treatment of consequences of CVI. | 6 hours
  The efficacy of using the ESVV for the treatment of deep CVI will be established by an increase of at least 100% in PPG recovery time (RT)

CONTACTS AND LOCATIONS:
Overall Officials: Arie Bass, Prof., Principal Investigator — Assaf Harofe Medical Center, Zrifin, Israel
Locations (1):
- Assaf Harofe Medical Center, Zrifin, Israel